CLINICAL TRIAL: NCT04892342
Title: An Open-Label, Multiple Dose, Dose Escalation and Cohort Expansion Phase I/II Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activities of ESG401 in Subjects With Locally Advanced/Metastatic Solid Tumors
Brief Title: Study of ESG401 in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Escugen Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ESG401-101
Record Dates: First submitted 2021-05-13; First posted 2021-05-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms, Breast; Neoplasms, Lung; Neoplasms,Colorectal; Neoplasms, Bladder; Neoplasm of Stomach; Neoplasms,Ovarian
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Stomach Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- ESG401 dose level 1 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 2 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 3 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 4 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 5 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 6 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 7 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 8 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 9 (Experimental)
  Interventions: Drug: ESG401
- ESG401 dose level 10 (Experimental)
  Interventions: Drug: ESG401

INTERVENTIONS:
Drug: ESG401 — Administered via intravenous (IV) infusion

SUMMARY:
The primary objective in Phase I is to evaluate the safety and tolerability of ESG401 as a single agent administered in 21-day treatment cycles in previously treated participants with advanced epithelial cancer. In Phase II, the primary objective is to evaluate the safety and efficacy of ESG401 administered in 21-day treatment cycles at a dose selected in Phase I.

Tumor types in the study will include: cervical, colorectal, endometrial, ovarian, esophageal, gastric adenocarcinoma, glioblastoma multiforme, head and neck cancers- squamous cell, hepatocellular, prostate, non-small-cell lung cancer, pancreatic, renal cell, small-cell lung cancer, non-triple negative breast cancer (non-TNBC), triple-negative breast cancer (TNBC) and metastatic urothelial cancer (mUC).

ELIGIBILITY:
Inclusion Criteria:

* Individuals able to understand and give written informed consent.
* Subjects must have a histologically or cytologically confirmed advanced or metastatic solid tumor(s) for which no effective standard therapy is available or tolerable.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* Subject must have adequate organ function
* Fertile men and women of childbearing potential must agree to use an effective method of birth control from providing signed consent and for 180 days after last investigational product administration. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause.

Exclusion Criteria:

* Subjects receiving cancer therapy (chemotherapy or other systemic anti-cancer therapies, immunotherapy, or radiation therapy) within 4 weeks before the first investigational product administration..
* Has not recovered from adverse events (e.g., returned to baseline or grade 0~1) due to a previously administered agent.

Note: Subjects with Grade 2 alopecia or anemia are exceptions to this criterion and may qualify for the study.

* Had major surgery within 4 weeks before dosing, or will not have fully recovered from surgery; or has surgery planned during the time the subject is expected to participate in the study or within 4 weeks after the last dose of study drug administration.
* Use of any investigational anti-cancer drug within 28 days before the first investigational product administration.
* New thromboembolic events, intestinal obstruction, gastrointestinal bleeding or perforation within 6 months
* Uncontrolled systemic bacterial, viral or fungal infections
* Subjects with symptomatic or untreated CNS metastases, or those requiring ongoing treatment for CNS metastases.
* Primary CNS malignancy; Or a second primary tumor other than the confirmed solid tumor within the previous 3 years
* Evidence of serious or uncontrolled systemic disease (e.g., unstable or decompensated respiratory disease, liver disease or kidney disease)
* Patients with gastrointestinal diseases (such as chronic gastritis, chronic enteritis or gastric ulcers), or with a previous history of severe or chronic diarrhea
* History of chronic skin disease and present skin disease (e.g. bullous dermatitis, acnelike rash, skin ulcer, etc.)
* Subjects with clinically significant cardiovascular disease as defined by the following:

  * Baseline left ventricular ejection fraction (LVEF) ≤ 50% measured by Echocardiogram (ECHO) or Multi-gated acquisition (MUGA)
  * Heart failure New York Heart Association (NYHA) Class II or above
  * Uncontrolled hypertension (BP ≥ 150/95 mmHg despite optimal therapy)
  * Prior or current cardiomyopathy
  * Atrial fibrillation with heart rate > 100 bpm
  * Unstable ischaemic heart disease (myocardial infarction (MI) within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly)
  * QTc interval >/= 450 msecs for male or >/= 470 msecs for female (Fridericia's formula: QTc=QT/RR0.33).
* Human Immunodeficiency Virus (HIV) infection.
* Subjects who are Hepatitis B surface antigen (HBsAg) and Hepatitis B core antibody (HBcAb) positive or Hepatitis C virus (HCV) antibody positive at screening must not be enrolled until further definite testing with Hepatitis B virus (HBV) DNA titres and HCV RNA tests can conclusively rule out presence of active infection (HBV DNA ≥ 1000 cps/mL or 200 IU/mL) requiring antiviral therapy with Hepatitis B and C, respectively
* Known immediate or delayed hypersensitivity reaction to irinotecan or other camptocampin derivatives such as topotecan or to have had grade ≥3 gastrointestinal reactions associated with irinotecan, or allergies, or to any investigational drug or excipient ingredient
* Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events and Serious Treatment Emergent Adverse Events | First dose date up to last dose plus 30 days
  Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) that begin or worsen on or after the start of study drug through 30 days after the last dose of study drug. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0. An AE that met one or more of the following outcomes was classified as serious:
  Fatal Life-threatening Disabling/incapacitating Results in hospitalization or prolongs a hospital stay A congenital abnormality Other important medical events may also be considered serious AEs if they may require medical or surgical intervention to prevent one of the outcomes listed above
Objective Response Rate (ORR) by Independent Central Review (ICR) | Up to 49 months
  ORR is defined as the rate an overall best response of either complete response (CR) or partial response (PR) by ICR assessment according to RECIST1.1. CR was defined as the disappearance of all target lesions and reduction in short axis of any pathologic lymphnode to <10 mm. PR was defined as ≥ 30% decrease in the sum of diameters of target lesions, taking the baseline sum diameters. Per planned analysis, ORR by ICR will be assessed for the TNBC Target Population in phase 2 only.

SECONDARY OUTCOMES:
Cmax | Up to 49 months
  Maximum observed plasma concentration
AUC0-inf | Up to 49 months
  Area under the serum concentration time curve from time 0 extrapolated to infinity
Objective Response Rate by Local Assessment | Up to 49 months
  ORR is defined as the rate an overall best response of either complete response (CR) or partial response (PR) by local assessment. CR was defined as the disappearance of all target lesions and reduction in short axis of any pathologic lymphnode to <10 mm. PR was defined as ≥3 0% decrease in the sum of diameters of target lesions, taking the baseline sum diameters. Per planned analysis, ORR by local assessment will be assessed for the Target Population both in phase 1 and phase 2.
Progression Free Survival (PFS) by Local Assessment | Up to 49 months
  Progression-free survival (PFS) is defined as the interval from the first dose start date to the date of disease progression defined as documented progressive disease (PD) or death from any cause, whichever occurs first.
Overall Survival by Local Assessment | Up to 49 months
  Overall survival is defined as the time from the date of the first dose start date to the date of death due to any cause.
ADA | Up to 49 months
  Incidence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Zhang Y, Bai R, Wu Y, Tong Z, Liu A, Zhang Y, Wang H, Wu X, Cheng Y, Yang H, Zhou Q, Xing X, Chen X, Qiu F, Ma F. Novel TROP2 antibody-drug conjugates for treatment of HER2-negative metastatic breast cancer patients with brain metastases: a promising option☆. ESMO Open. 2025 May;10(5):105059. doi: 10.1016/j.esmoop.2025.105059. Epub 2025 May 12. PMID 40359710
- [Derived] Wang J, Tong Z, Tan Y, Shi Y, Wu Y, Zhou Q, Xing X, Chen X, Qiu F, Ma F. Phase 1a study of ESG401, a Trop2 antibody-drug conjugate, in patients with locally advanced/metastatic solid tumors. Cell Rep Med. 2024 Sep 17;5(9):101707. doi: 10.1016/j.xcrm.2024.101707. Epub 2024 Aug 30. PMID 39216478